CLINICAL TRIAL: NCT00628823
Title: Treatment of Mild Enteropathy Celiac Disease
Acronym: TMCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Academy of Finland (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Kalle Kurppa, MD., PhD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SA-115376
Record Dates: First submitted 2008-02-24; First posted 2008-03-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Endomysial antibodies; Mild enteropathy; Treatment; Gluten-free diet
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (No Intervention): Gluten-containing diet
- A2 (Active Comparator): Gluten-free diet
  Interventions: Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: Gluten-free diet — Gluten containing foods removed from diet
  Other Names: No other names
  Arms: A2

SUMMARY:
The main purpose of this study is to evaluate the natural history of gluten sensitivity in endomysial antibody positive adults with celiac disease suspicion, who were found to have a only mild enteropathy (Marsh I-II) in the small-bowel mucosa. The investigators hypothesize that these subject are indeed gluten-sensitive, as measured by clinical, serological and histological indicators. If this would be the case, the current diagnostic criteria for celiac disease might need re-evaluation.

DETAILED DESCRIPTION:
The current diagnostic criteria of celiac disease require small-bowel mucosal villous atrophy with crypt hyperplasia (Marsh III). However, the mucosal damage develops gradually and the patients may have clinical symptoms and endomysial antibodies before the development of villous atrophy.

The main purpose of this study is to evaluate the natural history of gluten sensitivity in endomysial antibody positive adults with celiac disease suspicion, who were found to have a only mild enteropathy (Marsh I-II) in the small-bowel mucosa. We hypothesize that these subject are indeed gluten-sensitive, as measured by clinical, serological and histological indicators. If this would be the case, the current diagnostic criteria for celiac disease might need re-evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Celiac disease suspicion
* Positive endomysial antibodies
* At least Marsh I -type small-bowel mucosal lesion

Exclusion Criteria:

* Earlier celiac disease diagnosis
* Consuming oral corticosteroids or immune suppressants

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-03; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Small-Bowel mucosal morphology | one year

SECONDARY OUTCOMES:
Endomysial antibodies, tissue transglutaminase antibodies, Small-Bowel mucosal inflammation, clinical symptoms, laboratory parameters, bone mineral density. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Katri Kaukinen, MD, PhD, Principal Investigator — Tampere University
Locations (1):
- University of Tampere, Tampere, Finland